CLINICAL TRIAL: NCT00892164
Title: Thyroid Surgery With the New Harmonic Scalpel or the Electrothermal Bipolar Vessel Sealer: a Prospective Randomized Study
Brief Title: Thyroid Surgery With the New Harmonic Scalpel or the Electrothermal Bipolar Vessel Sealer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hippocration General Hospital (Other)
Responsible Party: Department of Endocrine Surgery, 1st Department of Propaedeutic Surgery, Hippocration General Hospital of Athens, Department of Endocrine Surgery, 1st Department of Propaedeutic Surgery, Hippocration General Hospital of Athens, Athens Medical School, University of Athens
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 642
Record Dates: First submitted 2009-04-30; First posted 2009-05-04 (Estimated); Last update posted 2009-05-04 (Estimated); Status verified 2009-05

CONDITIONS: Thyroidectomy
Keywords: thyroid surgery; total thyroidectomy; harmonic scalpel; electrothermal bipolar vessel sealer; hemostatic device

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- FOCUS (Group A) (Active Comparator): Patients submitted to total thyroidectomy with the use of the FOCUS harmonic scalpel device
  Interventions: Device: harmonic scalpel device (FOCUS)
- LIGASURE (Group Β) (Active Comparator): Patients submitted to total thyroidectomy with the use of the electrothermal bipolar vessel sealing device
  Interventions: Device: electrothermal bipolar vessel sealing system (LIGASURE PRECISE)

INTERVENTIONS:
Device: harmonic scalpel device (FOCUS) — hemostatic device utilized intraoperatively
  Arms: FOCUS (Group A)
Device: electrothermal bipolar vessel sealing system (LIGASURE PRECISE) — hemostatic device utilized intraoperatively
  Arms: LIGASURE (Group Β)

SUMMARY:
The objective of this study is to compare the results of total thyroidectomy using the new harmonic scalpel device to that with the electrothermal bipolar vessel sealer.

DETAILED DESCRIPTION:
The harmonic scalpel and the electrothermal bipolar vessel sealing system (LIGASURE PRECISE) have been both shown to be safe and effective in thyroid surgery. The moderate dissection capabilities of the previous harmonic scalpel instruments available for thyroid surgery have led to an innovative technical improvement of the device (FOCUS) that has very recently been implemented and has been made available in 2008. Comparison of the utilization of this new device, however, with the electrothermal bipolar vessel sealer has not been performed in any study. The objective of this study is to compare the results of total thyroidectomy using the FOCUS to that with the LIGASURE device in respect to hemostasis, operative time and perioperative complications. All patients undergoing a total thyroidectomy in our endocrine surgery department are randomized into those operated with FOCUS (Group A) and those with LIGASURE (Group B).

ELIGIBILITY:
Inclusion Criteria:

* total thyroidectomy

Exclusion Criteria:

* hemithyroidectomy or subtotal thyroidectomy
* additional surgical procedures together with the total thyroidectomy (i.e., parathyroidectomy or cervical lymph node dissection)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2008-08; Primary Completion 2008-12 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Hemostasis | intraoperatively (from skin incision to skin closure) & postoperatively (from skin closure until 1 week postoperatively)
Postoperative complications including laryngeal nerve palsy, hypocalcemia, hemorrhage, hematoma, wound infection and skin burn | postoperatively (from the day of surgery until 3-6 months postoperatively)
Operative time | from skin incision to skin closure

SECONDARY OUTCOMES:
Length of hospital stay | postoperatively (from the day of surgery until discharge)

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Manouras, MD, PhD, Principal Investigator — Department of Endocrine Surgery, 1st Department of Propaedeutic Surgery, Hippocration General Hospital of Athens, Athens Medical School, University of Athens, Athens, Greece
Locations (1):
- Department of Endocrine Surgery, 1st Department of Propaedeutic Surgery, Hippocration General Hospital of Athens, Athens Medical School, University of Athens, Athens, Abelokipoi (Vas. Sofias 114 Av.), Greece